CLINICAL TRIAL: NCT06970977
Title: CRS Questionnaire Validation Project
Status: Recruiting | Type: Observational
Sponsor: The European Forum for Research and Education in Allergy and Airway Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: S68027
Record Dates: First submitted 2025-04-15; First posted 2025-05-14 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Chronic Rhinosinusitis (CRS) With and Without Nasal Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The 'CRS validation project' consists of a joint effort of 32 medical centers in Europe, the USA, and South Africa to carry out the validation of 2 novel questionnaires designated to measure self-perceived severity and control of Chronic Rhinosinusitis (with or without nasal polyps).

This study will validate translated versions of the same set of questionnaires simultaneously in the centers involved after recruiting a total of 1000 patients, while data collection, statistical analysis, and creation of the study report will be carried out by the statistical department of the University of Leuven.

Patients will be recruited from the regular ENT practice of their hospital to minimize the complexity of the study.

DETAILED DESCRIPTION:
The objectives of this study are as follows:

* Validation of two new questionnaires with the aim of measuring the current perceived condition of a patient with chronic rhinosinusitis in terms of control and severity.
* Validation of these questionnaires in routine medical settings.
* Evaluation of the results of these questionnaires in comparison with other tools currently available.

ELIGIBILITY:
Inclusion Criteria:

* Patient capable of giving informed consent
* Diagnosis of chronic rhinosinusitis with or without nasal polyposis according to the EPOS guidelines
* No recent sinus surgery (within the last three months)

Exclusion Criteria:

* Not capable of giving informed consent
* No CRS
* Recent sinus surgery (within the last three months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, capable of giving consent, with certified CRS and no recent sinus surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Validation of a new questionnaire | Through study completion, an average of 6 months
  Validation of a questionnaire based on similar questionnaires already approved for use in other airway diseases. The aim to measure the current perceived status of a patient with chronic rhinosinusitis in terms of control and severity.
  A new questionnaire will be tested and compared with current tools. For this purpose, a set of questionnaires has been developed including the EPOS criteria for chronic rhinosinusitis, the SNOT-22, the patient global assessment tool and the VAS scores, among others.
  All these questionnaires will be completed by the patient at visit 1 and the results will be analysed once the recruitment target of 1,000 patients has been reached.
  No second patient participation is required.
Evaluation of the results | Through study completion, an average of 6 months
  Evaluation of the results of this questionnaire in comparison with other tools currently available.
  Once the target of recruiting 1000 patients has been reached, the results will be statistically analysed.
  Parallels will be drawn between the responses obtained by the usual means and those captured in the questionnaires to be validated.
  It is expected that, in all cases, the degree of control and severity represented in the questionnaires to be validated will conform to the EPOS criteria and to the results of the questionnaires usually used.
  The results will be compared for each of the new questionnaires in general and separately by language.
  The ultimate goal is to validate what will become the diagnostic gold standard for chronic rhinosinusitis.

SECONDARY OUTCOMES:
Validation of a new questionnaire | Through study completion, an average of 6 months
  Validation of a questionnaire based on feedback collected from patients with CRS where they expressed which are the symptoms that most afflict them or are most present, related to their disease. The aim to measure the current perceived status of a patient with chronic rhinosinusitis in terms of control and severity.
  A new questionnaire will be tested and compared with current tools. For this purpose, a set of questionnaires has been developed including the EPOS criteria for chronic rhinosinusitis, the SNOT-22, the patient global assessment tool and the VAS scores, among others.
  All these questionnaires will be completed by the patient at visit 1 and the results will be analysed once the recruitment target of 1,000 patients has been reached.
  No second patient participation is required.
Evaluation of the results | Through study completion, an average of 6 months
  Evaluation of the results of this questionnaire in comparison with other tools currently available.
  Once the target of recruiting 1000 patients has been reached, the results will be statistically analysed.
  Parallels will be drawn between the responses obtained by the usual means and those captured in the questionnaires to be validated.
  It is expected that, in all cases, the degree of control and severity represented in the questionnaires to be validated will conform to the EPOS criteria and to the results of the questionnaires usually used.

CONTACTS AND LOCATIONS:
Locations (32):
- United States (5):
  - UCLA Santa Monica Medical Center, Santa Monica, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Brigham Sinus Center at Brigham and Women's Hospital, Boston, Massachusetts
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Eastern Virginia Medical School, Virginia City, Virginia
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- St. Michael's Hospital, Toronto, Canada
- Univ of Copenhagen, Copenhagen, Denmark
- Germany (2):
  - HNO-Klinik, Universitätsklinikum Düsseldorf, Düsseldorf
  - Univ Munich, Munich
- Greece (2):
  - University General Hospital of Heraklion, Heraklion
  - U. Aristotle, Thessaloniki
- Univ Hospital Roma, Roma, Italy
- Netherlands (2):
  - Univ Amsterdam, Amsterdam
  - Alrijne Zorggroep, Leiden
- University of Oradea, Oradea, Romania
- Ahmed Alkhadi Hospital, Durban, South Africa
- Spain (14):
  - Hospital Clínico Universitario de Compostela, A Coruña
  - Hospital Clinic Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital de La Línea de La Concepción, Cadiz
  - Hospital Universitario Jerez de La Frontera, Cadiz
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Puerto Real, Cadiz
  - Hospital Universitario Fuenlabrada, Madrid
  - Hospital Universitario Infanta Elena, Madrid y Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital del Bierzo, Ponferrada
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital General Universitario de Valencia, Valencia